CLINICAL TRIAL: NCT00650650
Title: Comparison of Ultrasound Versus Radiography for Diagnosis of Nasal Fractures
Status: Completed | Type: Observational
Sponsor: Klinikum der Universitaet Muenchen, Grosshadern (Other)
Responsible Party: Robert Gürkov, MD, Klinikum der Universitaet Muenchen, Grosshadern
Other Study IDs: NF-US-XR-05
Record Dates: First submitted 2008-03-28; First posted 2008-04-02 (Estimated); Last update posted 2009-04-21 (Estimated); Status verified 2009-04

CONDITIONS: Nasal Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The standard imaging procedure to diagnose a nasal fracture still is radiography (lateral nasal view and occipitomental view). But technological advances in ultrasonography during the last few decades have made high-resolution ultrasound devices available to the majority of medical centers. It has been shown that the bony structures of the nose can be well examined by ultrasound in the last few years. The hypothesis: "Is ultrasound of equal diagnostic accuracy in diagnosing nasal fractures as radiography" is being tested in the investigators' study. Patients with suspected nasal fracture undergo ultrasound examination in addition to the routine x-ray imaging. After completion of treatment, the readings of both ultrasound and radiographs are compared in terms of sensitivity and specificity to diagnose nasal fractures.

ELIGIBILITY:
Inclusion Criteria:

* suspected nasal fracture

Exclusion Criteria:

* further fractures
* pregnancy
* unstable condition
* refusal to undergo ultrasound examination

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected nasal fracture.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik für Hals-Nasen-Ohrenheilkunde, LMU München, München, Bavaria, Germany